CLINICAL TRIAL: NCT00589914
Title: A Randomized, Double-Blind, Parallel-Group, Comparative Study of Flexible Doses of Paliperidone Palmitate and Flexible Doses of Risperidone Long-Acting Intramuscular Injection in Subjects With Schizophrenia
Brief Title: Comparison of Paliperidone Palmitate and RISPERDAL CONSTA in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012289; R092670PSY3006 (Other: Unique Protocol Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-10 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; long-acting injectable antipsychotic medication
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RISPERDAL CONSTA (Active Comparator): RISPERDAL CONSTA 25-50 mg eq every 2 weeks
  Interventions: Drug: RISPERDAL CONSTA
- R092670 (Experimental): Paliperidone Palmitate 50-150 mg eq every 4 wks
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: RISPERDAL CONSTA — RISPERDAL CONSTA: Type=exact number, unit=mg, number=25, 37.5, or 50, form=suspension for injection, route=Intramuscular use. One i.m. injection of RISPERDAL CONSTA 25-50 mg eq every 2 weeks at V4, V6, V7, V8, V9, and V10. PALIPERIDONE PALMITATE PLACEBO: Form=suspension for injection, route=Intramuscular use. One i.m. injection every 2 weeks at Baseline and at V4, V7, and V9. RISPERIDONE: Type=up to, unit=mg, number=1 to 6, form=Tablet, route=Oral Use. One tablet for the first 4 weeks (28 days) of the DB treatment period.
  Arms: RISPERDAL CONSTA
Drug: Paliperidone palmitate — PALIPERIDONE PALMITATE: Type=exact number, unit=mg, number=50, 100, or 150, form=suspension for injection, route=Intramuscular use. One i.m. injection of Paliperidone palmitate 50-150 mg eq every 4 wks at Baseline, V4, V7, and V9. RISPERDAL CONSTA PLACEBO: Form=suspension for injection, route=Intramuscular use. One i.m. injection every 4 weeks at Baseline, V4, V7, and V9.
  Arms: R092670

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of paliperidone palmitate in patients with Schizophrenia.

DETAILED DESCRIPTION:
This is a randomized (patients assigned to treatment groups by chance), double-blind (patient and study staff will not know the treatment assignment) study of paliperidone palmitate compared with RISPERDAL CONSTA (Risperidone Long-Acting Intramuscular Injection) in adult patients with schizophrenia. The total duration of the study will be approximately 14 weeks. For those patients without source documentation of tolerability to oral (by mouth) risperidone or paliperidone Extended Release (ER) tablets, injectable RISPERDAL CONSTA or paliperidone palmitate, or those patients who were not currently taking another antipsychotic, a minimum of 4 days and a maximum of 6 days of oral paliperidone ER treatment at a dosage of 6 mg/day will be administered for tolerability testing before the first injection of double-blind (DB) study drug (paliperidone palmitate or RISPERDAL CONSTA). During the DB period, study drug will be administered to patients as an intramuscular (i.m.) injection. Paliperidone palmitate (PP) 150mg equivalent (eq) (and RISPERDAL CONSTA placebo) at Baseline (BL) (Day 1), 100mg eq at Visit (V) 4 (Day 8), 50 or 100mg eq at V7 (Day 36), and 50,100,or 150mg eq at V9 (Day 64) or RISPERDAL CONSTA (RC) 25mg at V4 and V6 (Day 22), 25 or 37.5mg at V7, and 25, 37.5, or 50mg at V9 will be given as i.m. injections. Patients in the RC group will also take risperidone tablets (1-6 mg/day) at BL for 28 days and be given an injection of PP placebo at BL, V1, V7, and V9.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria as specified by the protocol for at least 1 year before screening
* Prior medical records, written documentation or verbal information obtained from previous psychiatric providers obtained by the investigator must be consistent with the diagnosis of schizophrenia
* A total PANSS score between 60 and 120, inclusive, at screening and baseline; Body mass index (BMI) at the screening visit BMI at least 17 kg/m2
* Female patients must be postmenopausal for at least 2 years, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before study entry and throughout the study as specified by the protocol. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (b hCG) pregnancy test result at screening.

Exclusion Criteria:

* Patient unable to provide consent or involuntarily committed to psychiatric hospitalization; A primary, active DSM-IV diagnosis on Axis I other than schizophrenia
* A DSM-IV diagnosis of active substance dependence within 3 months before screening (nicotine and caffeine are not exclusionary)
* History of treatment resistance as defined by failure to respond to 2 adequate treatments with different antipsychotic medications (an adequate treatment is defined as a minimum of 6 weeks at maximum tolerated dosage)
* Relevant history or current presence of any significant or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular disease), renal, hepatic, hematologic, endocrine, immunologic, or other systemic disease including history of neuroleptic malignant syndrome; History of any severe pre-existing gastrointestinal narrowing or inability to swallow oral study drug whole with the aid of water (applies to those patients requiring oral tolerability only)
* Significant risk of suicidal or violent behavior, as clinically assessed by the investigator ; History of life-threatening allergic reaction to any drug; Known or suspected hypersensitivity or intolerance to risperidone, paliperidone, 20% Intralipid, or any of their excipients (e.g., soybean oil, egg yolks, phospholipids, and glycerol)
* Have received an experimental drug or experimental biologic, or used an experimental medical device within 6 months before screening; History of any active malignancy within the previous 5 years, with the exception of basal cell carcinomas
* Women who are pregnant or breast-feeding or are planning to become pregnant uring the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1221 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (82):
- United States (15):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Cerritos, California
  - Garden Grove, California
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Flowood, Mississippi
  - Hollis, New York
  - Willoughby, Ohio
  - Oklahoma City, Oklahoma
  - DeSoto, Texas
  - Houston, Texas
  - Odessa, Texas
- Austria (3):
  - Linz
  - Salzburg
  - Vienna
- Bulgaria (2):
  - Plovdiv
  - Varna
- Czechia (6):
  - Brno
  - Dobřany
  - Kroměříž
  - Kutná Hora
  - Olomouc
  - Prague
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- France (3):
  - Bourges Cedex N/A
  - Dole
  - Romans-sur-Isère
- Germany (9):
  - Achim
  - Berlin
  - Bielefeld
  - Bochum
  - Jena
  - Leipzig
  - Mannheim
  - München
  - Stralsund
- Hungary (5):
  - Baja
  - Budapest
  - Gyõr
  - Kalocsa
  - Nagykálló
- India (6):
  - Aurangabad
  - Bangalore
  - Chandigarh
  - Mangalore
  - Pune
  - Varanasi
- Lithuania (4):
  - Alytus
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (10):
  - Bełchatów
  - Bytom Na
  - Chełmno
  - Gdynia Na
  - Katowice Woj Slaskie
  - Krakow Na
  - Lubliniec
  - Piekary Slaskie Na
  - Skorzewo Na
  - Warszawa Na
- Russia (6):
  - Moscow
  - Moscow Russia
  - Nizny Novgorod
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Spain (3):
  - Barcelona
  - Madrid
  - San Juan
- Ukraine (7):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Alphs L, Bossie CA, Fu DJ, Ma YW, Kern Sliwa J. Onset and persistence of efficacy by symptom domain with long-acting injectable paliperidone palmitate in patients with schizophrenia. Expert Opin Pharmacother. 2014 May;15(7):1029-42. doi: 10.1517/14656566.2014.909409. PMID 24754314
- [Derived] Fu DJ, Bossie CA, Sliwa JK, Ma YW, Alphs L. Paliperidone palmitate versus oral risperidone and risperidone long-acting injection in patients with recently diagnosed schizophrenia: a tolerability and efficacy comparison. Int Clin Psychopharmacol. 2014 Jan;29(1):45-55. doi: 10.1097/YIC.0000000000000006. PMID 24113628
- [Derived] Fu DJ, Bossie CA, Kern Sliwa J, Ma YW, Alphs L. Paliperidone palmitate versus risperidone long-acting injection in markedly-to-severely ill schizophrenia subjects: onset of efficacy with recommended initiation regimens. Clin Schizophr Relat Psychoses. 2014 Jul;8(2):101-9, 109A. PMID 23446197
- [Derived] Pandina G, Lane R, Gopal S, Gassmann-Mayer C, Hough D, Remmerie B, Simpson G. A double-blind study of paliperidone palmitate and risperidone long-acting injectable in adults with schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jan 15;35(1):218-26. doi: 10.1016/j.pnpbp.2010.11.008. Epub 2010 Nov 16. PMID 21092748
- See also: A Randomized, Double-Blind, Parallel-Group, Comparative Study of Flexible Doses of Paliperidone Palmitate and Flexible Doses of Risperidone Long-Acting Intramuscular Injection in Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=744&filename=CR012289_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 13 week double-blind study to assess safety and efficacy of flexible dose of Paliperidone Palmitate (50, 100 or 150 mg equivalent) in patients aged 18 years or older with schizophrenia.
Pre-assignment Details: In this study 1221 patients were enrolled of which 1220 patients were randomized as 1 patient was enrolled twice. Only the first patient number was included in the all randomized patients, safety, and intent to treat analysis sets. Out of 1220 patients 1214 patients received at least 1 dose of study medication.
Groups:
- R092670: Double-blind period. Flexible dose of 50, 100 or 150 mg equivalent administered by i.m. injection every 4 weeks up to Week 9 (Day 64).
- RISPERDAL CONSTA: Double-blind period. Flexible dose of 25, 37.5 or 50 mg administered by i.m. injection every 2 weeks up to Week 11 (Day 78).
Period: Overall Study
Arm/Group | R092670 | RISPERDAL CONSTA
Started | 606 | 608
Completed | 456 | 471
Not Completed | 150 | 137
Not completed — Adverse Event | 19 | 10
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 40 | 43
Not completed — Lost to Follow-up | 11 | 18
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 55 | 49
Not completed — Other | 22 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R092670 | RISPERDAL CONSTA | Total
Number analyzed (Participants) | 606 | 608 | 1214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 596 | 599 | 1195
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12.13) | 38.7 (11.83) | 38.9 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 268 | 513
  Male | 361 | 340 | 701
Region of Enrollment [Number; unit: participants]
  Austria | 3 | 3 | 6
  Bulgaria | 15 | 14 | 29
  Czech Republic | 50 | 48 | 98
  Estonia | 32 | 34 | 66
  France | 7 | 3 | 10
  Germany | 4 | 4 | 8
  Hungary | 31 | 34 | 65
  India | 31 | 31 | 62
  Lithuania | 17 | 20 | 37
  Poland | 24 | 20 | 44
  Russia | 159 | 159 | 318
  Spain | 17 | 17 | 34
  Ukraine | 84 | 84 | 168
  United States of America | 132 | 137 | 269
AgeCategorical [Number; unit: participants]
  18-25 years | 103 | 92 | 195
  26-50 years | 381 | 397 | 778
  51-65 years | 115 | 113 | 228
  >65 years | 7 | 6 | 13
  <18 years | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the Positive and Negative Syndrome Scale (PANSS) Total Score for Schizophrenia
Description: The PANSS scale is used to assess the neuropsychiatric symptoms of schizophrenia. The 30-item PANSS scale provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items),and the general psychopathology subscale (16 items), each item rated on a scale of 1 (absent) to 7 (extreme).
Time Frame: Baseline to the last postrandomization assessment in the double-blind treatment period (approximately 13 weeks)
Population: The per-protocol analysis set of patients included those randomized to treatment after IEC/ IRB approval of protocol Amendment INT-4 with both a baseline measurement and at least 1 postrandomization measurement on the primary efficacy variable, a minimum exposure of 36 days to the double-blind treatment regimen, and no major protocol violations.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | R092670 | RISPERDAL CONSTA
Number analyzed (Participants) | 389 | 376
Scores on a scale | -18.6 (15.45) | -17.9 (14.24)
Statistical Analysis 1: Comparison: R092670 vs RISPERDAL CONSTA; Null hypothesis: Difference between groups (RISPERDAL CONSTA minus paliperidone palmitate) for the mean change from baseline to endpoint in PANSS total score (LOCF) was less than or equal to -5 (prespecified non-inferiority margin). Sample size: SD of 20 for the change in PANSS total score, a true difference between treatment groups of 0.1 in favor of RISPERDAL CONSTA, 2-sided significance level of 5%, and 80% power. A sample size reestimation was performed when 60% of the data was available; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 5 points in the change in PANSS total score i.e., lower limit of the 95% CI for difference between groups (RISPERDAL CONSTA minus paliperidone palmitate) had to be greater than -5 to demonstrate non-inferiority; ANCOVA — No p-value to report; ANCOVA model with factors treatment, country and baseline score. Weighted approach used to account for interim analysis for sample size re-estimation; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.62 to 2.38], Standard Error of Mean 1.02

2. Secondary Outcome: The Change From Baseline for the CGI-S Score
Description: The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe). This scale permits a global evaluation of the patient's condition at a given time. A qualified rater administered the CGI-S.
Time Frame: Baseline to the last postrandomization assessment in the double-blind treatment period (approximately 13 weeks)]
Population: The intent-to-treat (ITT) analysis set of patients included those randomized to treatment after IEC/IRB approval of protocol Amendment INT-4 who received at least 1 injection of double-blind study drug and had at least 1 efficacy measurement during the double-blind treatment period.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | R092670 | RISPERDAL CONSTA
Number analyzed (Participants) | 453 | 460
Scores on a scale | -0.9 (0.97) | -0.9 (0.93)
Statistical Analysis 1: Comparison: R092670 vs RISPERDAL CONSTA; The change from baseline was analyzed using an ANCOVA model with factors for treatment and country and baseline score as a covariate; Test type: Superiority or Other; ANCOVA — No P-values reported; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.07 to 0.17], Standard Error of Mean 0.06

3. Secondary Outcome: The Change From Baseline in the PSP Score
Description: The PSP scale is used to assess the degree of dysfunction a patient exhibits over a 7-day period within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The results of the assessment are converted to a numeric score. A score between 71 and 100 indicates a mild degree of difficulty; a score between 31 and 70 indicates a moderate degree of dysfunction, and a patient with a score of 30 or less has functioning so poor he or she requires intensive supervision.
Time Frame: Baseline to the last postrandomization assessment in the double-blind treatment period (approximately 13 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | R092670 | RISPERDAL CONSTA
Number analyzed (Participants) | 448 | 452
Scores on a scale | 8.5 (11.82) | 8.8 (11.65)
Statistical Analysis 1: Comparison: R092670 vs RISPERDAL CONSTA; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA — No P-values reported; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.22 to 1.69], Standard Error of Mean 0.74

ADVERSE EVENTS:
Arm/Group | R092670 | RISPERDAL CONSTA
Serious Adverse Events (participants affected / at risk) | 41/606 | 29/608
Other Adverse Events (participants affected / at risk) | 147/606 | 108/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R092670 (N=606) | RISPERDAL CONSTA (N=608)
Constipation (Gastrointestinal disorders) | 0 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 3 | 1
Psychotic disorder (Psychiatric disorders) | 13 | 7
Schizophrenia (Psychiatric disorders) | 15 | 13
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Tension (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R092670 (N=606) | RISPERDAL CONSTA (N=608)
Injection site pain (General disorders) | 31 | 5
Headache (Nervous system disorders) | 43 | 44
Somnolence (Nervous system disorders) | 34 | 24
Insomnia (Psychiatric disorders) | 57 | 41

LIMITATIONS AND CAVEATS:
Of 1221 patients randomized, one patient was enrolled twice and assigned 2 patient numbers. Only the first patient number is included in the results reported for 1220 randomized patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days